CLINICAL TRIAL: NCT02400788
Title: A Phase I/II Study in Combination of Resminostat and Sorafenib in Patients With Advanced Hepatocellular Carcinoma Previously Untreated With Systemic Chemotherapy
Brief Title: Resminostat (YHI-1001) in Combination With Sorafenib in Asian Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YHI-1001-HCC-02
Record Dates: First submitted 2015-03-10; First posted 2015-03-27 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — resminostat; Sorafenib

ARMS (2):
- Resminostat + Sorafenib (Experimental): oral administration
  Interventions: Drug: Resminostat; Drug: Sorafenib
- Sorafenib (Active Comparator): oral administration
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Resminostat
  Arms: Resminostat + Sorafenib
Drug: Sorafenib

SUMMARY:
The purpose of this study is to assess efficacy and safety in combination of resminostat and sorafenib in Asian patients with advanced HCC previously untreated with systemic chemotherapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with advanced or metastatic hepatocellular carcinoma
* Patients with ECOG PS of 0-1
* Patients who can be treated with oral medications and have no gastrointestinal function disorder which is considered to affect the absorption of medications

Main Exclusion Criteria:

* Patients with a history of treatment with HDAC inhibitors
* Pregnant women and lactating mothers
* Patients with brain metastases or suspected brain metastases based on the clinical symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2013-04; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Phase 1 : Number of participants with dose limited toxicities as measure of safety and tolerability | 6 months
Phase 2 : Time To Progression (TTP) | 12 months

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (9):
  - Chiba
  - Ishikawa
  - Kanagawa
  - Kochi
  - Kyoto
  - Osaka
  - Saga
  - Shizuoka
  - Tokyo
- South Korea (3):
  - Busan
  - Daegu
  - Seoul